CLINICAL TRIAL: NCT01214148
Title: A Prospective, Multi-centre, Single Treatment Clinical Trial With Follow-up Investigations at 1, 4, 9, 12, 24 and 36 Months
Brief Title: First in Man Experience With a Drug Eluting Stent in De Novo Coronary Artery Lesions
Acronym: BIOFLOW-I
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Biotronik AG (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: C0904
Record Dates: First submitted 2010-09-30; First posted 2010-10-04 (Estimated); Last update posted 2013-08-12 (Estimated); Status verified 2013-08

CONDITIONS: Coronary Artery Disease
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- ORSIRO (Other)
  Interventions: Device: ORSIRO - Drug Eluting Coronary Stent

INTERVENTIONS:
Device: ORSIRO - Drug Eluting Coronary Stent — The coronary stent is delivered to the intended implantation location by means of the fast-exchange delivery system and then expanded to its final diameter by dilating the balloon. It remains in the vessel as a permanent implant.

SUMMARY:
A prospective, single-treatment, multi centre clinical trial enrolling 30 patients in 2 centres in Romania, with a clinical and angiographic follow-up at 4 and 9 months to determine the primary endpoint of late lumen loss and secondary endpoints. A subgroup of 15 patients will also undergo post implantation, 4 and 9 months IVUS examinations. Additional clinical follow-ups take place at 1 month and yearly up to three (3) years.

The objective of this trial is to assess the safety and clinical performance of the ORSIRO drug eluting stent in patients with single de-novo coronary artery lesions.

ELIGIBILITY:
Inclusion Criteria:

1. Patient is ≥18 years old;
2. Clinical evidence of ischemic heart disease and / or a positive functional study. Documented stable angina pectoris (Canadian cardiovascular society classification (CCS) 1, 2, 3 or 4 ), or documented silent ischemia;
3. Single de novo lesion with ≥50% and <90% stenosis in 1 coronary artery;

Exclusion Criteria:

1. Documented left ventricular ejection fraction (LVEF) ≤30%;
2. Unstable angina pectoris(Braunwald Class A I-III)
3. Three-vessel coronary artery disease
4. Evidence of myocardial infarction within 72 hours prior to the index procedure;
5. Known allergies to the following: Acetylsalicylic acid (ASA) (Aspirin®), Clopidogrel bisulfate (Plavix®.) or Ticlopidine (Ticlid®.), Heparin, contrast agent (that cannot be adequately premedicated), cobalt-chromium (CoCr), Poly-L-Lactidic Acid (PLLA), silicon carbide (aSiC:H)
6. A platelet count <100.000 cells/mm3 or >700.000 cells/mm3 or a WBC <3.000 cells/mm3;
7. Acute or chronic renal dysfunction (serum creatinine >2.0 mg/dl or >150µmol/L);
8. Total occlusion (TIMI 0 or 1);
9. Target vessel has evidence of thrombus or is excessively tortuous that makes it unsuitable for proper stent delivery and deployment;
10. Significant (>50%) stenosis proximal or distal to the target lesion that might require revascularization or impede run off;
11. Heavily calcified lesion and/or calcified lesion which cannot be successfully predilated;
12. Target lesion is located in or supplied by an arterial or venous bypass graft;
13. Ostial target lesion (within 5.0mm of vessel origin);
14. Target lesion involves a side branch >2.0mm in diameter;
15. Unprotected Left main coronary artery disease (stenosis >50%);

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2009-07; Primary Completion 2010-04 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
In-stent Late Lumen Loss | 9 months post procedure

SECONDARY OUTCOMES:
In-stent and in-segment binary restenosis rate | 4 and 9 months post procedure.
In-stent and in-segment (proximal and distal) minimum lumen diameter | 4 and 9 months post-procedure
In-segment late lumen loss | 4 and 9 months post procedure
In-stent late lumen loss | 4 months post procedure.
Target Lesion Revascularization | 1, 4 and 9 months and at 1, 2 and 3 years post-procedure
Clinically driven target lesion revascularization | 1, 4 and 9 months and at 1, 2 and 3 years post-procedure
Target Vessel Revascularization | 1, 4 and 9 months and at 1, 2 and 3 years post-procedure
- Composite of cardiac death, MI attributed to the target vessel and clinically driven target lesion revascularization | 1, 4 and 9 month post-procedure, and yearly up to 3 years
- Composite of all-cause mortality, any MI and any revascularization, target vessel revascularization or revascularization of nontarget vessels | 3 years post procedure
Stent thrombosis | 1, 4 and 9 months and 1, 2 and 3 years post-procedure
Neointimal hyperplasia volume (subgroup) | 4 and 9 months post-procedure measured by Intravascular Ultrasound (IVUS)

CONTACTS AND LOCATIONS:
Overall Officials: Martial Hamon, MD, Principal Investigator — Centre Hospitalier Universitaire Caen
Locations (2):
- Romania (2):
  - Institutul de Urgenţă pentru Boli Cardiovasculare "Prof. Dr. C. C. Iliescu" - Spitalul Clinic Fundeni, Bucharest
  - Spitalul Clinic de Urgenţă Bucureşti, Bucharest